CLINICAL TRIAL: NCT02584257
Title: Comparison of the Pharmacodynamic Profile of Test and Reference Metered Dose Inhalers (MDIs) Containing Albuterol Sulfate Using Bronchoprovocation in Adult Patients With Stable Mild Asthma
Brief Title: Pharmacodynamic Bioequivalence of Metered Dose Inhalers of Albuterol Sulfate in Patients With Stable Mild Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lupin, Inc. (Industry)
Responsible Party: Sponsor
Organization: Lupin Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AS-MDI-301
Record Dates: First submitted 2015-10-12; First posted 2015-10-22 (Estimated); Results first posted 2020-11-18 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Mild Persistent Asthma
MeSH Terms: interventions — Methacholine Chloride; Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo dose (Placebo Comparator): Placebo dose: 1 actuation each from 2 different placebo ProAir HFA inhalation aerosols and one actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols
  Interventions: Other: methacholine chloride; Drug: placebo ProAir HFA; Drug: placebo Lupin albuterol HFA MDI
- 90 mcg ProAir HFA (Active Comparator): 90 mcg of ProAir HFA: 1 actuation each from ProAir HFA inhalation aerosol and the placebo ProAir HFA inhalation aerosol and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols
  Interventions: Other: methacholine chloride; Drug: placebo ProAir HFA; Drug: ProAir HFA; Drug: placebo Lupin albuterol HFA MDI
- 180 mcg ProAir HFA (Active Comparator): 180 mcg of ProAir HFA: 1 actuation each from 2 different ProAir HFA inhalation aerosols and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols
  Interventions: Other: methacholine chloride; Drug: ProAir HFA; Drug: placebo Lupin albuterol HFA MDI
- 90 mcg Lupin albuterol HFA MDI (Experimental): 90 mcg of Lupin albuterol HFA MDI product: 1 actuation each from the Lupin albuterol HFA MDI inhalation aerosol and the placebo Lupin albuterol HFA MDI inhalation aerosol and 1 actuation each from 2 different placebo ProAir HFA inhalation aerosols
  Interventions: Other: methacholine chloride; Drug: placebo ProAir HFA; Drug: Lupin albuterol HFA MDI; Drug: placebo Lupin albuterol HFA MDI
- 180 mcg Lupin albuterol HFA MDI (Experimental): 180 mcg of Lupin albuterol HFA MDI: 1 actuation each from 2 different Lupin albuterol HFA MDI inhalation aerosols and 1 actuation each from 2 different placebo ProAir HFA product inhalation aerosols
  Interventions: Other: methacholine chloride; Drug: placebo ProAir HFA; Drug: Lupin albuterol HFA MDI

INTERVENTIONS:
Other: methacholine chloride
Drug: placebo ProAir HFA
  Arms: 180 mcg Lupin albuterol HFA MDI; 90 mcg Lupin albuterol HFA MDI; 90 mcg ProAir HFA; Placebo dose
Drug: ProAir HFA
  Arms: 180 mcg ProAir HFA; 90 mcg ProAir HFA
Drug: Lupin albuterol HFA MDI
  Arms: 180 mcg Lupin albuterol HFA MDI; 90 mcg Lupin albuterol HFA MDI
Drug: placebo Lupin albuterol HFA MDI
  Arms: 180 mcg ProAir HFA; 90 mcg Lupin albuterol HFA MDI; 90 mcg ProAir HFA; Placebo dose

SUMMARY:
The purpose of this study is to demonstrate the pharmacodynamic bioequivalence of the test product to the reference product, using bronchoprovocation (methacholine challenge testing) in adult patients with stable mild asthma.

DETAILED DESCRIPTION:
A Multicenter, Double-Blind, Double-Dummy, Placebo-Controlled, 5-Treatment, Randomized, Crossover Study to Demonstrate the Pharmacodynamic Bioequivalence of Test and Reference Metered Dose Inhalers containing Albuterol Sulfate using Bronchoprovocation in Adult Patients with Stable Mild Asthma

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female subjects (18-65 years of age)
* Stable mild asthmatics based on National Asthma Education and Prevention Program (NAEPP) guidelines.
* Forced Expiratory Volume in 1 second ( FEV1) ≥ 80% of predicted. Airway responsiveness to methacholine demonstrated by a pre-albuterol dose (baseline) PC20 ≤ 8 mg/ml.
* Nonsmokers for at least 1 year prior to the study and a maximum smoking history of five pack-years (the equivalent of one pack per day for five years).
* Written informed consent.

Exclusion Criteria:

* Conditions which could alter airway reactivity to methacholine (e.g., pneumonia, upper respiratory tract infection, lower respiratory tract, viral bronchitis and/or sinobronchitis) within six weeks preceding the screening visit.
* History of seasonal asthma exacerbations, in which case the patient should be studied outside of the relevant allergen season.
* History of cystic fibrosis, bronchiectasis or other respiratory diseases.
* History of cardiovascular, renal, neurologic, liver or endocrine dysfunction, or chronic condition that could put the safety of the patient at risk during the study or affect the efficacy and safety analyses during the study.
* Treatment in an emergency room, urgent care center, or hospitalization for acute asthmatic symptoms within the past 6 months or need for daily oral corticosteroids within past 3 months.
* Known intolerance or hypersensitivity to any component of the albuterol metered dose inhaler (MDI).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2016-04; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Investigational Research Center Site #110, Huntington Beach, California
  - Investigational Research Center Site #114, Mission Viejo, California
  - Investigational Research Center Site #113, Rolling Hills Estates, California
  - Investigational Research Center Site #112, San Diego, California
  - Investigational Research Center Site #116, San Jose, California
  - Investigational Research Center Site #106, Tallahassee, Florida
  - Investigational Research Center Site #109, Baltimore, Maryland
  - Investigational Research Center Site #105, Bethesda, Maryland
  - Investigational Research Center Site #103, North Dartmouth, Massachusetts
  - Investigational Research Center Site #108, St Louis, Missouri
  - Investigational Research Center Site #115, Bellevue, Nebraska
  - Investigational Research Center Site #104, Skillman, New Jersey
  - Investigational Research Center Site #102, Raleigh, North Carolina
  - Investigational Research Center Site #111, Cincinnati, Ohio
  - Investigational Research Center Site #118, Tulsa, Oklahoma
  - Investigational Research Center Site #101, Medford, Oregon
  - Investigational Research Center Site #107, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male/female patients 18-65 years of age, inclusive, with a diagnosis of asthma and at least a 6-month history of stable mild asthma as defined by the NAEPP EPR-3 guidelines were recruited and enrolled at 17 different centers in the USA. First subject was screened on April 12th, 2016 and the last patient was completed the study on August 12th, 2016.
Pre-assignment Details: Of the 217 patients enrolled in the study, 126 failed screening or were randomization failures, largely due to failure to meet the inclusion and exclusion criteria. 91 Subjects were randomized to treatment groups.
Groups:
- PBO-R90-T180-R180-T90: Subjects received PBO in period 1 (1 actuation each from 2 different placebo ProAir HFA inhalation aerosols and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols), R90 in period 2 (1 actuation each from ProAir HFA inhalation aerosol and the placebo ProAir HFA inhalation aerosol and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols), T180 in period 3 (1 actuation each from 2 different Lupin albuterol HFA MDI inhalation aerosols and 1 actuation each from 2 different placebo ProAir HFA product inhalation aerosols), R180 in period 4 (1 actuation each from 2 different ProAir HFA inhalation aerosols and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols), T90 in period 5 (1 actuation each from the Lupin albuterol HFA MDI inhalation aerosol and the placebo Lupin albuterol HFA MDI inhalation aerosol and 1 actuation each from 2 different placebo ProAir HFA inhalation aerosols)
- R90-R180-PBO-T90-T180: Subjects received R90 in period 1 (1 actuation each from tProAir HFA inhalation aerosol and the placebo ProAir HFA inhalation aerosol and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols), R180 in period 2 (1 actuation each from 2 different ProAir HFA inhalation aerosols and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols), PBO in period 3 (1 actuation each from 2 different placebo ProAir HFA inhalation aerosols and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols), T90 in period 4 (1 actuation each from the Lupin albuterol HFA MDI inhalation aerosol and the placebo Lupin albuterol HFA MDI inhalation aerosol and 1 actuation each from 2 different placebo ProAir HFA inhalation aerosols), T180 in period 5 (1 actuation each from 2 different Lupin albuterol HFA MDI inhalation aerosols and 1 actuation each from 2 different placebo ProAir HFA product inhalation aerosols)
- R180-T90-R90-T180-PBO: Subjects received R180 in period 1 (1 actuation each from 2 different ProAir HFA inhalation aerosols and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols), T90 in period 2 (1 actuation each from the Lupin albuterol HFA MDI inhalation aerosol and the placebo Lupin albuterol HFA MDI inhalation aerosol and 1 actuation each from 2 different placebo ProAir HFA inhalation aerosols), R90 in period 3 (1 actuation each from ProAir HFA inhalation aerosol and the placebo ProAir HFA inhalation aerosol and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols), T180 in period 4 (1 actuation each from 2 different Lupin albuterol HFA MDI inhalation aerosols and 1 actuation each from 2 different placebo ProAir HFA product inhalation aerosols), PBO in period 5 (1 actuation each from 2 different placebo ProAir HFA inhalation aerosols and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols)
- T90-T180-R180-PBO-R90: Subjects received T90 in period 1 (1 actuation each from the Lupin albuterol HFA MDI inhalation aerosol and the placebo Lupin albuterol HFA MDI inhalation aerosol and 1 actuation each from 2 different placebo ProAir HFA inhalation aerosols), T180 in period 2 (1 actuation each from 2 different Lupin albuterol HFA MDI inhalation aerosols and 1 actuation each from 2 different placebo ProAir HFA product inhalation aerosols), R180 in period 3 (1 actuation each from 2 different ProAir HFA inhalation aerosols and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols), PBO in period 4 (1 actuation each from 2 different placebo ProAir HFA inhalation aerosols and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols), R90 in period 5 (1 actuation each from tProAir HFA inhalation aerosol and the placebo ProAir HFA inhalation aerosol and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols)
- T180-PBO-T90-R90-R180: Subjects received T180 in period 1 (1 actuation each from 2 different Lupin albuterol HFA MDI inhalation aerosols and 1 actuation each from 2 different placebo ProAir HFA product inhalation aerosols), PBO in period 2 (1 actuation each from 2 different placebo ProAir HFA inhalation aerosols and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols), T90 in period 3 (1 actuation each from the Lupin albuterol HFA MDI inhalation aerosol and the placebo Lupin albuterol HFA MDI inhalation aerosol and 1 actuation each from 2 different placebo ProAir HFA inhalation aerosols), R90 in period 4 (1 actuation each from tProAir HFA inhalation aerosol and the placebo ProAir HFA inhalation aerosol and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols), R180 in period 5 (1 actuation each from 2 different ProAir HFA inhalation aerosols and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols)
- T90-R180-T180-R90-PBO: Subjects received T90 in period 1 (1 actuation each from the Lupin albuterol HFA MDI inhalation aerosol and the placebo Lupin albuterol HFA MDI inhalation aerosol and 1 actuation each from 2 different placebo ProAir HFA inhalation aerosols), R180 in period 2 (1 actuation each from 2 different ProAir HFA inhalation aerosols and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols), T180 in period 3 (1 actuation each from 2 different Lupin albuterol HFA MDI inhalation aerosols and 1 actuation each from 2 different placebo ProAir HFA product inhalation aerosols), R90 in period 4 (1 actuation each from tProAir HFA inhalation aerosol and the placebo ProAir HFA inhalation aerosol and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols), PBO in period 5 (1 actuation each from 2 different placebo ProAir HFA inhalation aerosols and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols)
- T180-T90-PBO-R180-R90: Subjects received T180 in period 1 (1 actuation each from 2 different Lupin albuterol HFA MDI inhalation aerosols and 1 actuation each from 2 different placebo ProAir HFA product inhalation aerosols), T90 in period 2 (1 actuation each from the Lupin albuterol HFA MDI inhalation aerosol and the placebo Lupin albuterol HFA MDI inhalation aerosol and 1 actuation each from 2 different placebo ProAir HFA inhalation aerosols), PBO in period 3 (1 actuation each from 2 different placebo ProAir HFA inhalation aerosols and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols), R180 in period 4 (1 actuation each from 2 different ProAir HFA inhalation aerosols and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols), R90 in period 5 (1 actuation each from tProAir HFA inhalation aerosol and the placebo ProAir HFA inhalation aerosol and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols)
- R90-PBO-R180-T180-T90: Subjects received R90 in period 1 (1 actuation each from tProAir HFA inhalation aerosol and the placebo ProAir HFA inhalation aerosol and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols), PBO in period 2 (1 actuation each from 2 different placebo ProAir HFA inhalation aerosols and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols), R180 in period 3 (1 actuation each from 2 different ProAir HFA inhalation aerosols and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols), T180 in period 4 (1 actuation each from 2 different Lupin albuterol HFA MDI inhalation aerosols and 1 actuation each from 2 different placebo ProAir HFA product inhalation aerosols), T90 in period 5 (1 actuation each from the Lupin albuterol HFA MDI inhalation aerosol and the placebo Lupin albuterol HFA MDI inhalation aerosol and 1 actuation each from 2 different placebo ProAir HFA inhalation aerosols)
- R180-R90-T90-PBO-T180: Subjects received R180 in period 1 (1 actuation each from 2 different ProAir HFA inhalation aerosols and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols), R90 in period 2 (1 actuation each from tProAir HFA inhalation aerosol and the placebo ProAir HFA inhalation aerosol and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols), T90 in period 3 (1 actuation each from the Lupin albuterol HFA MDI inhalation aerosol and the placebo Lupin albuterol HFA MDI inhalation aerosol and 1 actuation each from 2 different placebo ProAir HFA inhalation aerosols), PBO in period 4 (1 actuation each from 2 different placebo ProAir HFA inhalation aerosols and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols), T180 in period 5 (1 actuation each from 2 different Lupin albuterol HFA MDI inhalation aerosols and 1 actuation each from 2 different placebo ProAir HFA product inhalation aerosols),
Period: Period 1
Arm/Group | PBO-R90-T180-R180-T90 | R90-R180-PBO-T90-T180 | R180-T90-R90-T180-PBO | T90-T180-R180-PBO-R90 | T180-PBO-T90-R90-R180 | T90-R180-T180-R90-PBO | T180-T90-PBO-R180-R90 | R90-PBO-R180-T180-T90 | R180-R90-T90-PBO-T180
Started | 9 | 9 | 9 | 8 | 10 | 10 | 18 | 9 | 9
Completed | 9 | 9 | 9 | 8 | 10 | 10 | 17 | 9 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Period 2
Arm/Group | PBO-R90-T180-R180-T90 | R90-R180-PBO-T90-T180 | R180-T90-R90-T180-PBO | T90-T180-R180-PBO-R90 | T180-PBO-T90-R90-R180 | T90-R180-T180-R90-PBO | T180-T90-PBO-R180-R90 | R90-PBO-R180-T180-T90 | R180-R90-T90-PBO-T180
Started | 9 | 9 | 9 | 8 | 10 | 10 | 17 | 9 | 9
Completed | 8 | 8 | 9 | 8 | 10 | 10 | 17 | 9 | 9
Not Completed | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | PBO-R90-T180-R180-T90 | R90-R180-PBO-T90-T180 | R180-T90-R90-T180-PBO | T90-T180-R180-PBO-R90 | T180-PBO-T90-R90-R180 | T90-R180-T180-R90-PBO | T180-T90-PBO-R180-R90 | R90-PBO-R180-T180-T90 | R180-R90-T90-PBO-T180
Started | 8 | 8 | 9 | 8 | 10 | 10 | 17 | 9 | 9
Completed | 8 | 8 | 9 | 8 | 10 | 10 | 17 | 9 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | PBO-R90-T180-R180-T90 | R90-R180-PBO-T90-T180 | R180-T90-R90-T180-PBO | T90-T180-R180-PBO-R90 | T180-PBO-T90-R90-R180 | T90-R180-T180-R90-PBO | T180-T90-PBO-R180-R90 | R90-PBO-R180-T180-T90 | R180-R90-T90-PBO-T180
Started | 8 | 8 | 9 | 8 | 10 | 10 | 17 | 9 | 9
Completed | 8 | 8 | 9 | 8 | 10 | 10 | 17 | 9 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | PBO-R90-T180-R180-T90 | R90-R180-PBO-T90-T180 | R180-T90-R90-T180-PBO | T90-T180-R180-PBO-R90 | T180-PBO-T90-R90-R180 | T90-R180-T180-R90-PBO | T180-T90-PBO-R180-R90 | R90-PBO-R180-T180-T90 | R180-R90-T90-PBO-T180
Started | 8 | 8 | 9 | 8 | 10 | 10 | 17 | 9 | 9
Completed | 8 | 8 | 9 | 8 | 10 | 10 | 17 | 9 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized patients who received a dose of any of the study medications.
Groups:
- Safety Population: All randomized patients who received a dose of any of the randomized study medications. Patient baseline characteristics are not designated by treatment arms due to the crossover design of the study (treatment groups are not mutually exclusive).
Arm/Group | Safety Population
Number analyzed (Participants) | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 91
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (11.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 63
  Black/African American | 25
  Asian | 1
  American Indian/Alaska Native | 0
  Native Hawaiian/Other Pacific Islander | 0
  Other | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 3
  Not Hispanic/Latino | 88
Region of Enrollment [Number; unit: participants] — The study was conducted in 17 study centers in the United States of America (USA)
  participants
    United States | 91

OUTCOME MEASURES:

1. Primary Outcome: Post-dose PC20 Concentration After Receiving Differing Doses of Test, Reference, or Placebo
Description: The primary efficacy endpoint was the postdose PC20 following administration of differing doses of albuterol (or placebo) by inhalation. The 20% reduction in FEV1 was determined relative to the saline stage FEV1 measured before albuterol or placebo administration. Additionally, an analysis of superiority to placebo was performed for the T and R products prior to the BE determination. In this study the ITT and PP populations were identical.
Time Frame: Post-dose at Visits 2-6 of the study, a total of approximately 4 weeks.
Population: Intent-to-Treat population included all randomized patients who completed at least 2 treatment periods with valid PC20 FEV1 measurements.Treatment was assigned based upon treatment to which patients had been randomized regardless of which treatment they actually received. This was primary population for comparisons of T and R products to placebo.
Measure: Least Squares Mean (Standard Error); unit: log(mg/mL)
Groups:
- Placebo Dose: Placebo dose: 1 actuation each from 2 different placebo ProAir HFA inhalation aerosols and one actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols
  methacholine chloride
  placebo ProAir HFA
  placebo Lupin albuterol HFA MDI N=82
- 90 mcg ProAir HFA: 90 mcg of ProAir HFA: 1 actuation each from ProAir HFA inhalation aerosol and the placebo ProAir HFA inhalation aerosol and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols
  methacholine chloride
  placebo ProAir HFA
  ProAir HFA
  placebo Lupin albuterol HFA MDI
- 180 mcg ProAir HFA: 180 mcg of ProAir HFA: 1 actuation each from 2 different ProAir HFA inhalation aerosols and 1 actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols
  methacholine chloride
  ProAir HFA
  placebo Lupin albuterol HFA MDI
- 90 mcg Lupin Albuterol HFA MDI: 90 mcg of Lupin albuterol HFA MDI product: 1 actuation each from the Lupin albuterol HFA MDI inhalation aerosol and the placebo Lupin albuterol HFA MDI inhalation aerosol and 1 actuation each from 2 different placebo ProAir HFA inhalation aerosols
  methacholine chloride
  placebo ProAir HFA
  Lupin albuterol HFA MDI
  placebo Lupin albuterol HFA MDI
- 180 mcg Lupin Albuterol HFA MDI: 180 mcg of Lupin albuterol HFA MDI: 1 actuation each from 2 different Lupin albuterol HFA MDI inhalation aerosols and 1 actuation each from 2 different placebo ProAir HFA product inhalation aerosols
  methacholine chloride
  placebo ProAir HFA
  Lupin albuterol HFA MDI
Arm/Group | Placebo Dose | 90 mcg ProAir HFA | 180 mcg ProAir HFA | 90 mcg Lupin Albuterol HFA MDI | 180 mcg Lupin Albuterol HFA MDI
Number analyzed (Participants) | 82 | 83 | 83 | 80 | 81
log(mg/mL) | 0.608 (0.239) | 3.779 (0.238) | 4.432 (0.238) | 3.928 (0.241) | 4.481 (0.240)
Statistical Analysis 1: Comparison: Placebo Dose vs 90 mcg ProAir HFA; Test type: Superiority; p < 0.0001, Brief Mixed Models Analysis — Fixed effects of dose, week, and sequence and the random effect of the patient was carried out to ensure that the overall treatment effect was significant at p<0.05; For this model, the dependent variable was log2(PC20FEV1) values where PC20FEV1 was measured in mg/mL; Least Square Means Differences = 3.171, 95% CI 2-sided [2.732 to 3.610], Standard Error of Mean 0.238
Statistical Analysis 2: Comparison: Placebo Dose vs 180 mcg ProAir HFA; Test type: Superiority; p < 0.0001, Brief Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; For this model, the dependent variable was log2(PC20FEV1) values where PC20FEV1 was measured in mg/mL; Least Square Means Differences = 3.824, 95% CI 2-sided [3.384 to 4.263], Standard Error of Mean 0.238
Statistical Analysis 3: Comparison: Placebo Dose vs 90 mcg Lupin Albuterol HFA MDI; Test type: Superiority; p < 0.0001, Brief Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; For this model, the dependent variable was log2(PC20FEV1) values where PC20FEV1 was measured in mg/mL; Least Square Means Differences = 3.320, 95% CI 2-sided [2.876 to 3.764], Standard Error of Mean 0.241
Statistical Analysis 4: Comparison: Placebo Dose vs 180 mcg Lupin Albuterol HFA MDI; Test type: Superiority; p < 0.0001, Brief Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; For this model, the dependent variable was log2(PC20FEV1) values where PC20FEV1 was measured in mg/mL; Least Square Means Differences = 3.872, 95% CI 2-sided [3.430 to 4.315], Standard Error of Mean 0.240
Statistical Analysis 5: Comparison: 90 mcg ProAir HFA vs 180 mcg ProAir HFA vs 90 mcg Lupin Albuterol HFA MDI vs 180 mcg Lupin Albuterol HFA MDI; An Emax model was developed and the 90% confidence interval of Frel was a bias corrected accelerated confidence interval based on a bootstrapping procedure. The bootstrapping procedure used for this analysis was residual resampling. The Per-Protocol population was the primary population for bioequivalence analysis. Patients in the PP population must have completed at least 2 treatment periods with valid PC20FEV1 measurements and had no major protocol deviations within those intervals; Test type: Equivalence — A blinded interim analysis was performed after 60 patients completed all treatment visits which determined that 80 subjects would be sufficient to complete the study with 90% power; Frel = 1.15, 90% CI 2-sided [0.93 to 1.48], Standard Error of Mean 0.17 — Frel is the relative bioavailability of the test versus reference product. The CI was a bias corrected and accelerated CI based on a bootstrapping procedure. The FDA acceptable CI was between 0.67 and 1.50

ADVERSE EVENTS:
Time Frame: All AE/SAEs (including treatment-emergent AEs) were assessed throughout the study visits and followed to resolution/satisfaction. AEs were recorded starting after the patient had signed the informed consent form and assessed at all visits. Each AE was evaluated for date/time of onset, duration, intensity, and causal relationship with the investigational product or other factors. (5 months) First Patient Screened: 12-Apr 2016 & Last Patient Visit: 12 Aug 2016
Description: An AE was defined as any untoward medical occurrence in a clinical trial patient administered a medicinal product and which did not necessarily have a causal relationship with the treatment. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational medicinal product, whether or not considered related to the investigational medicinal product.
Groups:
- Placebo Dose: Placebo dose: 1 actuation each from 2 different placebo ProAir HFA inhalation aerosols and one actuation each from 2 different placebo Lupin albuterol HFA MDI inhalation aerosols
  methacholine chloride
  placebo ProAir HFA
  placebo Lupin albuterol HFA MDI
Arm/Group | Placebo Dose | 90 mcg ProAir HFA | 180 mcg ProAir HFA | 90 mcg Lupin Albuterol HFA MDI | 180 mcg Lupin Albuterol HFA MDI
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/90 | 0/89 | 0/88 | 0/89
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/90 | 0/89 | 0/88 | 0/89
Other Adverse Events (participants affected / at risk) | 3/89 | 4/90 | 1/89 | 8/88 | 1/89
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Dose (N=89) | 90 mcg ProAir HFA (N=90) | 180 mcg ProAir HFA (N=89) | 90 mcg Lupin Albuterol HFA MDI (N=88) | 180 mcg Lupin Albuterol HFA MDI (N=89)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart Rate Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tension Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes